CLINICAL TRIAL: NCT00714493
Title: A Phase 4, Multicenter, Open-Label, Assessor-Blinded Switch Study of the Efficacy and Safety of Infliximab (REMICADE) in Patients With Active Rheumatoid Arthritis Who Are Responding Inadequately to Etanercept (ENBREL) or Adalimumab (HUMIRA).
Brief Title: RESTART C0168Z05 Rheumatoid Arthritis Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013879; C0168Z05 (Other: Centocor Ortho Biotech Services, L.L.C.); NCT01281449 (obsolete NCT alias)
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; remicade; infliximab; Centocor; etanercept; enbrel; adalimumab; humira; restart; swollen joints; tender joints.
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Other): Infliximab3 mg/kg at week 0,2,6; Increase to 5mg/kg or 7 mg/kg based on EULAR response
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — 3 mg/kg at week 0,2,6; Increase to 5mg/kg or 7 mg/kg based on EULAR response

SUMMARY:
The purpose of this study is to assess the effectiveness of treatment in patients with active rheumatoid arthritis who are having an inadequate response to at least 3 months of treatment with etanercept or adalimumab in addition to methotrexate.

DETAILED DESCRIPTION:
This is a Phase 4, multi center, open-label, assessor blinded, switch study of infliximab in patients with active rheumatoid arthritis who are receiving methotrexate and are having an inadequate response to their current treatment with etanercept or adalimumab. The last dose of etanercept must have been at least 1 week but not more than 2 weeks prior to the first infliximab study infusion. The last dose of adalimumab must have been administered at least 2 weeks but not more than 4 weeks prior to the first infliximab study infusion. The study will be conducted for 30 weeks and will include 200 patients. All eligible patients will receive 3 mg/kg infliximab infusions (drug given into a vein) at weeks 0, 2, and 6 and every 8 weeks thereafter, if they achieve a European League Against Rheumatism (EULAR) response on their current dose of infliximab. Patients who do not achieve a EULAR response will increase their dose from 3mg/kg to 5 mg/kg at week 14. Patients who do not achieve a EULAR response at week 22 will increase from either 3 mg/kg to 5 mg/kg or from 5mg/kg to 7 mg/kg. The last study infusion will take place at week 22. The last study visit for effectiveness evaluations will take place at week 26. A week 30 follow-up visit will be performed for adverse events and tuberculosis evaluations, health economics assessments, and review of concomitant medications. All patients who end the study early will be required to complete all assessments. Patients will receive 3 mg/kg infliximab infusions at weeks 0, 2, and 6. If patients achieve European League Against Rheumatism (EULAR) response, they will remain on their current dose. Patients who do not demonstrate a EULAR response will increase their infliximab dose from 3 mg/kg to 5 mg/kg at week 14. At week 22, patients will also increase their infliximab dose from 3 mg/kg to 5mg/kg or from 5 mg/kg to 7mg/kg if they do not demonstrate a EULAR response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have rheumatoid arthritis
* Patients must have greater than or equal to 6 tender joints and greater than or equal to 6 swollen joints
* Patients must have inadequate disease response to etanercept or adalimumab
* Patients must have received etanercept or adalimumab in combination with methotrexate for a minimum of at least 3 months prior to the screening visit. The last dose of etanercept must have been given at least 1 week but not more than 2 weeks prior to first infliximab infusion. The last dose of adalimumab must have been administered at least 2 weeks but not more than 4 weeks prior to first infliximab infusion.

Exclusion Criteria:

* Patients who have a history of latent or active TB
* Have inflammatory disease other than rheumatoid arthritis
* Have had a chronic or recurrent infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.
Locations (76):
- United States (45):
  - Huntsville, Alabama
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Santa Monica, California
  - Bridgeport, Connecticut
  - Lewes, Delaware
  - Boca Raton, Florida
  - Palm Harbor, Florida
  - Tamarac, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Moline, Illinois
  - Springfield, Illinois
  - Lexington, Kentucky
  - Wheaton, Maryland
  - Saint Clair Shores, Michigan
  - Eagan, Minnesota
  - Springfield, Missouri
  - St Louis, Missouri
  - Berkeley Heights, New Jersey
  - Freehold, New Jersey
  - Albany, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Mayfield, Ohio
  - Middleburg Heights, Ohio
  - Tulsa, Oklahoma
  - Allentown, Pennsylvania
  - Duncansville, Pennsylvania
  - Wexford, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Mesquite, Texas
  - Temple, Texas
  - Tyler, Texas
  - Burke, Virginia
  - Reston, Virginia
  - Seattle, Washington
- Austria (2):
  - Graz-Eggenberg
  - Vienna
- Canada (5):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Toronto, Ontario
  - Hamilton Ontario
- Helsinki, Finland
- France (4):
  - Bordeaux
  - Limoges
  - Montivilliers
  - Orléans
- Germany (5):
  - Frankfurt
  - Holdenfelde
  - Leipzig
  - München
  - Ratingen
- Israel (7):
  - Ashkelon
  - Beer Yaakov
  - Haifa
  - Kfar Saba
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Alkmaar, Netherlands
- Spain (3):
  - Madrid
  - Oviedo
  - Santiago de Compostela
- United Kingdom (3):
  - Leeds
  - London
  - Wigan

REFERENCES:
- [Derived] Fleischmann R, Goldman JA, Leirisalo-Repo M, Zanetakis E, El-Kadi H, Kellner H, Bolce R, DeHoratius R, Wang J, Decktor D. Infliximab efficacy in rheumatoid arthritis after an inadequate response to etanercept or adalimumab: results of a target-driven active switch study. Curr Med Res Opin. 2014 Nov;30(11):2139-49. doi: 10.1185/03007995.2014.942416. Epub 2014 Jul 30. PMID 25050591

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Infliximab 3 mg/kg (intravenously) at weeks 0,2,6; Increase to 5 mg/kg (i.v.) or 7 mg/kg (i.v.) based on EULAR response
Period: Overall Study
Arm/Group | Infliximab
Started | 203
Completed | 154
Not Completed | 49
Not completed — Adverse Event | 11
Not completed — Death | 3
Not completed — Lack of Efficacy | 10
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 12
Not completed — SUBJECT CHOICE (SUBJECT WITHDREW CONSENT | 8
Not completed — OTHER | 2

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 171
  >=65 years | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 42
Region of Enrollment [Number; unit: participants]
  Europe | 43
  North America | 160

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Achieved a EULAR (The European League Against Rheumatism) Response at Week 10
Description: Percent of patients who achieved EULAR response at Week 10. EULAR response is defined based on the DAS28 score and the EULAR response criteria (Van Gestel et al, 1996 and 1999). At a given visit, patients with a DAS28 score of ≤ 5.1 are considered EULAR responders if the improvement from baseline in their DAS28 score is greater than 0.6; Or patients with a DAS28 score > 5.1 are considered EULAR responders if the improvement from baseline in their DAS28 score is > 1.2.
Time Frame: Week 10
Population: The evaluable population was the subset of the mITT population (included the enrolled patients who received at least 1 dose of study medication) after excluding all 6 patients from Site 8631 where significant trial misconducts were identified.
Measure: Number; unit: Percentage
Groups:
- Infliximab 3 mg/kg: Infliximab 3 mg/kg at week 0,2,6; Increase to 5mg/kg or 7 mg/kg based on EULAR response
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 197
Percentage | 49.7 [42.6 to 56.9]

2. Secondary Outcome: Percent of Patients Who Acheived EULAR Response at Week 10 and Maintained Through Week 26 Without Infliximab Dose Increase
Description: Percent of patients who achieved EULAR response at Week 10 and maintained through Week 26 without infliximab dose increase
Time Frame: Week 26
Measure: Number; unit: percentage
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 197
percentage | 22.3 [16.7 to 28.8]

3. Secondary Outcome: Percent of Patients Who Achieved EULAR Response at Week 26, Regardless of EULAR Response Status at Weeks 10, 14, and 22, With or Without Dose Increase Prior to Week 26
Description: Percent of patients who achieved EULAR response at Week 26, regardless of EULAR response status at Weeks 10, 14, and 22, with or without dose increase prior to Week 26
Time Frame: Week 26
Measure: Number; unit: percentage
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 197
percentage | 51.8 [44.6 to 58.9]

4. Secondary Outcome: Change From Baseline in Physical Function (HAQ)
Description: Change from baseline in physical function (HAQ) at Week 10. HAQ assesses the degree of difficulty a person has in accomplishing tasks. A lower HAQ score indicates less difficulty. Change from baseline is computed as Week 10 value minus baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: scale -3 to 3
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 173
scale -3 to 3 | -0.173 (0.4548)
Statistical Analysis 1: Comparison: Infliximab 3 mg/kg; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; change from baseline

5. Secondary Outcome: Change From Baseline in Physical Function (HAQ)
Description: Change from baseline in physical function (HAQ) at Week 26. HAQ assesses the degree of difficulty a person has in accomplishing tasks. A lower HAQ score indicates less difficulty. Change from baseline is computed as Week 26 value minus baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Week 26
Measure: Mean (Standard Deviation); unit: scale -3 to 3
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 151
scale -3 to 3 | -0.223 (0.4968)
Statistical Analysis 1: Comparison: Infliximab 3 mg/kg; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test

6. Secondary Outcome: Percent of Patients Who Achieved ACR20 at Week 10
Description: Percent of patients who achieved ACR20 at Week 10. A patient is considered achieving ACR20 if the following two conditions are met: 1) An improvement of ≥ 20% from baseline in both the swollen joint count (66 joints) and tender joint count (68 joints; 2) An improvement of ≥ 20% from baseline in at least 3 of the following 5 assessments:Patient's assessment of pain visual analog scale (VAS), Patient's global assessment of disease activity (VAS), Evaluator's global assessment of disease activity (VAS), Patient's assessment of physical function as measured by the HAQ disability index, and CRP.
Time Frame: Week 10
Measure: Number; unit: percentage
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 197
percentage | 28.4 [22.2 to 35.3]

7. Secondary Outcome: Percent of Patients Who Achieved ACR20 at Weeks 26.
Description: Percent of patients who achieved ACR20 at Weeks 26. A patient is considered achieving ACR20 if the following two conditions are met: 1) An improvement of ≥ 20% from baseline in both the swollen joint count (66 joints) and tender joint count (68 joints; 2) An improvement of ≥ 20% from baseline in at least 3 of the following 5 assessments:Patient's assessment of pain visual analog scale (VAS), Patient's global assessment of disease activity (VAS), Evaluator's global assessment of disease activity (VAS), Patient's assessment of physical function as measured by the HAQ disability index, and CRP.
Time Frame: Week 26
Measure: Number; unit: percentage
Arm/Group | Infliximab 3 mg/kg
Number analyzed (Participants) | 197
percentage | 35.5 [28.9 to 42.7]

ADVERSE EVENTS:
Time Frame: All untoward events occurring between the time of obtaining informed consent through Week 30 or early termination were collected, regardless of causality.
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 10/203
Other Adverse Events (participants affected / at risk) | 54/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=203)
Cardiac Failure Congestive (Cardiac disorders) | 2
Acute Myocardial Infarction (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Atrioventricular Block Complete (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 1
Congestive Cardiomyopathy (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Multi-Organ Failure (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Erysipelas (Infections and infestations) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Completed Suicide (Psychiatric disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=203)
Sinusitis (Infections and infestations) | 17
Upper Respiratory Tract Infection (Infections and infestations) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Headache (Nervous system disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days